CLINICAL TRIAL: NCT07084662
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Xinlikang Capsule in the Treatment of Chemotherapy-induced Fatigue and Immune Disorders in Patients With Diffuse Large B Lymphoma
Brief Title: Xinlikang Capsule for Chemotherapy-induced Fatigue and Immune Disorders in Diffuse Large B Lymphoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, MD. PhD., Sun Yet-Sen University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2025-004
Record Dates: First submitted 2025-07-09; First posted 2025-07-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tebufenozide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xinlikang capsules (Experimental): The experimental group was treated with Xinlikang capsules after meals, 5 capsules each time, 3 times a day for 12 weeks.
  Interventions: Drug: Xinlikang capsules
- Mimic capsules (Placebo Comparator): The control group was treated with mimic capsules, 5 capsules each time after meals, 3 times a day for 12 weeks.
  Interventions: Drug: mimic capsules

INTERVENTIONS:
Drug: Xinlikang capsules — Xinlikang capsules after meals, 5 capsules each time, 3 times a day for 12 weeks
  Arms: Xinlikang capsules
Drug: mimic capsules — mimic capsules, 5 capsules each time after meals, 3 times a day for 12 weeks.
  Arms: Mimic capsules

SUMMARY:
To evaluate the efficacy and safety of Xinlikang capsule in the treatment of cancer-related fatigue (CRF) and peripheral blood lymphocytes in patients with diffuse large B-cell lymphoma (DLBCL) who achieved complete remission (CR) after all courses of chemotherapy-containing regimens

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Newly diagnosed diffuse large B lymphoma (DLBCL);
3. Patients had completed the first-line treatment of chemotherapy and immunotherapy and the course of treatment had been completed.
4. Metabolic complete response (CR) was evaluated by PET/CT during or after chemotherapy.
5. Had completed the full course of chemotherapy-containing regimen for more than 30-90 days;
6. BFI fatigue score ≥4;
7. The expected survival time was ≥6 months;
8. No treatment plan for CD20 monoclonal antibody, radiotherapy, chemotherapy, lenalidomide, thymopeptides, targeted drugs, biological agents, immunosuppressive agents, other Chinese medicine decoction or Chinese patent medicine in the next 3 months;
9. No grade 3-4 surgery plan is expected in the next 3 months;
10. They had normal mental consciousness, could understand the content of the questionnaire correctly, and could complete the questionnaire with assistance or independently;
11. Women and men of childbearing age agreed to use contraception during and for 1 month after treatment;
12. They volunteered to participate in the clinical trial and signed the informed consent form, which was in accordance with the requirements of Good Clinical Practice (GCP).

Exclusion Criteria:

1. DLBCL subjects with CNS involvement at initial diagnosis;
2. Allergic or intolerant to Xinlikang capsule or its component drugs;
3. Significant abnormal liver and kidney function: ALT, AST, GGT≥3 ULN; BUN and Cr≥3 ULN;
4. Severe abnormal bone marrow function: white blood cell ≤1.0×10^9/L, neutrophil ≤0.5×10^9/L, platelet ≤30×10^9/L, hemoglobin ≤6g/dL;
5. Patients with HIV virus infection, bacterial infection and other immune-related diseases that affect immune function as judged by clinicians;
6. Uncontrolled HBV or HCV infection: Hepatitis B Virus (HBV) DNA testing exceeding the lower limit of detection or 1000 copies /mL or 500 IU/mL (the higher is the reference) during screening in patients with a history of chronic hepatitis B; HCV RNA detection in patients with a history of Hepatitis C Virus (HCV) infection during the screening period exceeded the detection limit of the assay or 1000 copies /mL or 500 IU/mL (whichever was higher was used as a reference).
7. Patients with other malignancies.
8. Enrollment in another clinical trial 30 days before screening or during the trial;
9. Persons who were deemed by the investigator to be ineligible to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
The difference of FACIT Fatigue Scale score | From baseline to 12 weeks of treatment
  The scale ranges from 0 to 4, with lower scores indicating better outcomes.

SECONDARY OUTCOMES:
The difference of FACIT Fatigue Scale scores | Differences in FACIT Fatigue Scale scores from baseline at the end of 2, 4, and 8 weeks of treatment.
  The scale ranges from 0 to 4, with lower scores indicating better outcomes.
BFI | BFI differences from baseline at 2 weeks, 4 weeks, 8 weeks and 12 weeks of treatment
  The scale ranges from 0 to 10, with lower scores indicating better outcomes.
FACT-Lym total score | FACT-Lym total score differences from baseline at 2 weeks, 4 weeks, 8 weeks and 12 weeks of treatment
  The scale ranges from 0 to 4, with lower scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No